CLINICAL TRIAL: NCT04750837
Title: Autologous Platelet-Rich Plasma Versus Conventional Dressing Method in the Treatment of Chronic Diabetic Foot Ulcers
Brief Title: Platelet Rich Plasma and Diabetic Foot Ulcer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Yasser Ali Orban, principal investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Platelet rich plasma
Record Dates: First submitted 2021-02-07; First posted 2021-02-11 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Platelet Rich Plasma

STUDY DESIGN:
Intervention Model Description: 2 groups one group managed by conventional dressing and the other by platelet rich plasma
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet rich plasma group (Active Comparator): chronic diabetic foot ulcer was treated by platelet rich plasma
  Interventions: Procedure: debridement of the wound; Biological: platelet rich plasma; Procedure: conventional dressing
- conventional dressing group (Sham Comparator): chronic diabetic foot ulcer was treated by conventional dressing
  Interventions: Procedure: debridement of the wound; Procedure: conventional dressing

INTERVENTIONS:
Procedure: debridement of the wound — The edges and the floor of the wound were firstly debrided, and any callosities around the wound were removed. This was repeated if needed when callosities around the wound reappeared. By this technique, the chronic wound was transformed into an acute one
Biological: platelet rich plasma — Part of activated PRP was injected around the wound and under the base of the wound, while another portion of PRP was left over the floor of the wound and let to coagulate and form a gel.
  Arms: Platelet rich plasma group
Procedure: conventional dressing — The wound was irrigated by normal saline, covered by vaseline gauze then sterile dressing. Repeated dressing every two days till 20 weeks, if the wound failed to heal at that time

SUMMARY:
In chronic diabetic foot ulcer, if the conventional dressing fails, new therapeutic options such as recombinant human growth factors and bioengineered skin substitutes may be beneficial, but the cost is a limiting factor. Autologous platelet rich plasma is a cost-effective method that enhances wound healing by promoting the healing process by local release of growth factors.

DETAILED DESCRIPTION:
The term "chronic wound" was first used in literature in the 1950s to refer to wounds that were difficult to heal or did not follow a normal healing process. However, the term has met criticism for its uncertainty regarding the duration of chronicity. Martin & Nunan, 2015, defined a "chronic wound" as a barrier defect that has not healed in 3 months, and Leaper & Durani, 2008, defined it as a wound that lacks a 20-40% reduction in its size after 2-4 weeks of optimal treatment or when there is no complete healing after 6 weeks. Recent reviews have highlighted the lack of consensus regarding the definition of a "chronic wound" and the need for further researches in this area.

Diabetic foot ulcer is a major complication of diabetes mellitus and is the major component of diabetic foot syndrome. This medical condition affects 15% of all patients with diabetes mellitus. Alvarsson et al. in 2012 reported that up to 88% of all lower leg amputations were related to diabetic foot ulcers.

The impact of chronic wounds on the health and quality of patients' life and their families should not be underestimated. Patients with chronic wounds may experience chronic pain, loss of function and mobility, depression, and anxiety, increased social stress and isolation, prolonged hospitalization, increased financial burden, and increased morbidity and mortality.

Growth factors (GFs) play an essential role in the process of wound healing and tissue regeneration. Each GF has more than one effect on the healing process and acts by binding to specific cell membrane receptors on the target cells. Growth factors' effects include promoting chemotaxis, inducing cell migration and proliferation, and stimulate cells to upregulate protein production. These growth factors not only regulate cell migration and proliferation but also promote angiogenesis and remodel the extracellular matrix, creating an ideal environment that favors the cutaneous wound healing process.

Over the last decades, the use of emerging cellular therapies, such as platelet-rich plasma (PRP), has more attention in a variety of diseases and settings for its potential use in the regenerative medicine as a therapeutic agent and can have an adjunctive role in a standardized, quality treatment plan.

PRP is defined as plasma containing above-baseline concentrations of platelets, which is from 140 000-400 000/μl. PRP is isolated through the centrifugation of whole blood. Simply, its actions are based on the infusion of elevated platelets, thereby theoretically enhancing the biological healing capacity and tissue generation in the wound bed. Enzyme-linked immunosorbent assay studies of PRP have quantified the presence of increases in GFs such as transforming GF β, epidermal GF, and platelet-derived GF. Through degranulation of the alpha granules in platelets, PRP can secrete various GFs, which have been documented to initiate the wound healing process

ELIGIBILITY:
Inclusion Criteria:

- Patients with chronic diabetic foot ulcers more than 1 cm in diameter that failed to heal in three months after wound debridement and dressing by a surgeon.

Exclusion Criteria:

1. Patients with evident local infection or gangrene (no redness, no hotness, no purulent discharge, no osteomyelitis in X-ray with a negative probe to bone test, and negative C-reactive protein).
2. Patients with end-stage organ failure, hepatic, or renal failure.
3. Patients on anticoagulants.
4. Patients on antiplatelet agents.
5. Patients with thrombocytopenia.
6. Patients on steroid therapy.
7. Ulcers less than 1cm or greater than 8 cm in diameter.
8. Deep ulcers more than 2 cm in depth.
9. Patients with lower limb ischemia (acute or chronic). Limb ischemia was excluded by the detection of the distal limb pulsations with ankle-brachial index>0.9.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2020-01-16 (Actual); Primary Completion 2020-12-21 (Actual); Study Completion 2021-01-20 (Actual)

PRIMARY OUTCOMES:
size of the ulcer reduce to zero cm | 20 weeks
  complete coverage of the ulcer base by healthy tissue

CONTACTS AND LOCATIONS:
Overall Officials: Yasser A. Orban, Lecturer, Principal Investigator — zagazig university faculty of human medicine
Locations (1):
- Zagazig University Faculty of Human Medicine, Zagazig, Sharqia Province, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] GREELEY PW. Plastic surgical closure of chronic open wounds of the leg. Ind Med Surg. 1953 Jan;22(1):22-3. No abstract available. PMID 13022118
- [Background] CARLESON R, GARSTEN P. [Wound therapy with septofyllin, with special consideration of its effect on chronic leg ulcers]. Nord Med. 1952 Mar 28;47(13):412-6. No abstract available. Undetermined Language. PMID 14941406
- [Background] Martin P, Nunan R. Cellular and molecular mechanisms of repair in acute and chronic wound healing. Br J Dermatol. 2015 Aug;173(2):370-8. doi: 10.1111/bjd.13954. Epub 2015 Jul 14. PMID 26175283
- [Background] Leaper DJ, Durani P. Topical antimicrobial therapy of chronic wounds healing by secondary intention using iodine products. Int Wound J. 2008 Jun;5(2):361-8. doi: 10.1111/j.1742-481X.2007.00406.x. PMID 18494641
- [Background] Gould L, Abadir P, Brem H, Carter M, Conner-Kerr T, Davidson J, DiPietro L, Falanga V, Fife C, Gardner S, Grice E, Harmon J, Hazzard WR, High KP, Houghton P, Jacobson N, Kirsner RS, Kovacs EJ, Margolis D, McFarland Horne F, Reed MJ, Sullivan DH, Thom S, Tomic-Canic M, Walston J, Whitney J, Williams J, Zieman S, Schmader K. Chronic wound repair and healing in older adults: current status and future research. Wound Repair Regen. 2015 Jan-Feb;23(1):1-13. doi: 10.1111/wrr.12245. Epub 2015 Feb 13. PMID 25486905
- [Background] Baba M, Davis WA, Norman PE, Davis TM. Temporal changes in the prevalence and associates of foot ulceration in type 2 diabetes: the Fremantle Diabetes Study. J Diabetes Complications. 2015 Apr;29(3):356-61. doi: 10.1016/j.jdiacomp.2015.01.008. Epub 2015 Jan 19. PMID 25670409
- [Background] Jarbrink K, Ni G, Sonnergren H, Schmidtchen A, Pang C, Bajpai R, Car J. Prevalence and incidence of chronic wounds and related complications: a protocol for a systematic review. Syst Rev. 2016 Sep 8;5(1):152. doi: 10.1186/s13643-016-0329-y. PMID 27609108